CLINICAL TRIAL: NCT01174719
Title: Phase 4 Study Comparing Albumin 5%, Hydroxyethylstrach 130/0.4 (6%) and Ringer Lactate for Volume Replacement During Cardiac Surgery
Brief Title: Humanalbumin, Hydroxyethylstarch and Ringer Lactate During Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Eva M. Base, Associate Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HAHes
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Valvular Heart Disease; Coronary Artery Disease
Keywords: Hydroxyethylstarch; Humanalbumin; Ringer Lactate; patients undergoing cardiac surgery
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease | interventions — HES 130-0.4; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hydroxyethylstarch (Active Comparator)
  Interventions: Drug: volume replacement
- Humanalbumin (Active Comparator)
  Interventions: Drug: Humanalbumin 5%
- Ringer lactate (Active Comparator)
  Interventions: Drug: volume replacement

INTERVENTIONS:
Drug: volume replacement — Hydroxyethylstarch up to 50mL/kg/24 hrs
  Other Names: Voluven; HES 130/0.4
  Arms: Hydroxyethylstarch
Drug: Humanalbumin 5% — Humanalbumin 5% up to 50 mL/kg/24 hours
  Other Names: Humanalbumin 5% Baxter
  Arms: Humanalbumin
Drug: volume replacement — up 10 50mL/kg/24 hours
  Arms: Ringer lactate

SUMMARY:
The aim of the study is to compare three different regimens for volume replacement during cardiac surgery, e.g. Albumin 5%, Hydroxyethylstarch 130/0.4 (HES) and Ringer-Lactate (RL).

Main Outcome parameters: chest tube drainage and coagulation parameters. The investigators hypothesis is that HES is as safe as Albumin, however less expensive. Whether RL is an even less expensive and as safe alternative has to be shown.

ELIGIBILITY:
Inclusion Criteria:

* Valve replacement
* Coronary bypass surgery

Exclusion Criteria:

* Severe left ventricular dysfunction
* Coagulation disorders

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-03; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
chest tube drainage | 24 hours

SECONDARY OUTCOMES:
Hemoglobin concentration | induction of anesthesia = baseline
Hematocrit value | induction of anesthesia = baseline
platelet count | induction of anesthesia = baseline
activated clotting time | induction of anesthesia = baseline
Modified thromboelastometry coagulation analysis (ROTEM, Pentapharm, Munich, Germany) | induction of anethesia = baseline
  using 3 activators: intrinsic ROTEM (InTEM, extrinsic ROTEM (ExTEM), finbrinogen ROTEM (FibTEM)
Hemoglobin concentration | average 1 hour on cardiopulmonary bypass
Hematocrit value | average 1 hour on cardiopulmonary bypass
Modified thromboelastometry coagulation analysis (ROTEM, Pentapharm, Munich, Germany) | average 1 hour on cardiopulmonary bypass
  using 3 activators: intrinsic ROTEM (InTEM, extrinsic ROTEM (ExTEM), finbrinogen ROTEM (FibTEM)
activated clotting time | average 1 hour on cardiopulmonary bypass
Hemoglobin concentration | 30 minutes after arrival ICU
Hematocrit value | 30 minutes after arrival ICU
platelet count | 30 minutes after arrival ICU
activated clotting time | 30 minutes after arrival ICU
Modified thromboelastometry coagulation analysis (ROTEM, Pentapharm, Munich, Germany) | 30 minutes after arrival ICU
  using 3 activators: intrinsic ROTEM (InTEM, extrinsic ROTEM (ExTEM), finbrinogen ROTEM (FibTEM)
Hemoglobin concentration | 24 hours after surgery
Hematocrit value | 24 hours after surgery
platelet count | 24 hrs after surgery
Modified thromboelastometry coagulation analysis (ROTEM, Pentapharm, Munich, Germany) | 24 hrs after surgery
  using 3 activators: intrinsic ROTEM (InTEM, extrinsic ROTEM (ExTEM), finbrinogen ROTEM (FibTEM)

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Base, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Vienna General Hospital, Vienna, Vienna, Austria